CLINICAL TRIAL: NCT02308592
Title: Patient Decision Aid (PDA) for Antidepressant Use In Pregnancy
Brief Title: Patient Decision Aid for Antidepressant Use in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Simone Vigod, Psychiatrist, Women's College Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Pregnancy; Depression
Keywords: Pregnancy; Depression; Antidepressant Use; Decision Aid
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Resource Sheet (Placebo Comparator): Women allocated to the control intervention will login to the study website and receive a printable PDF containing references to standard published information on antidepressant use in pregnancy. This ensures women have access to accurate information on the benefits and risks of antidepressant medication in pregnancy (even though they will not receive the PDA).
  Interventions: Behavioral: Standard Resource Sheet
- Electronic Patient Decision Aid (Active Comparator): The electronic Patient Decision Aid (PDA) is an interactive website with 3 main sections:
  1. Evidence-based information on (a) depression in pregnancy, (b) each treatment option and procedure;
  2. (a) Evidence-based information on the risks and benefits of both untreated depression and antidepressant treatment, (b) exercises to help women determine which risks and benefits are most important to them; and
  3. A summary section that outlines the information reviewed and which benefits and risks they deemed most important.
  At the end of the PDA, women allocated to this intervention will ALSO receive the standard resource sheet which is being used as the placebo comparator.
  Interventions: Behavioral: Electronic Patient Decision Aid; Behavioral: Standard Resource Sheet

INTERVENTIONS:
Behavioral: Electronic Patient Decision Aid — The electronic Patient Decision Aid (PDA) is an interactive website with 3 main sections:
  1. Evidence-based information on (a) depression in pregnancy, (b) each treatment option and procedure;
  2. (a) Evidence-based information on the risks and benefits of both untreated depression and antidepressant treatment, (b) exercises to help women determine which risks and benefits are most important to them; and
  3. A summary section that outlines the information reviewed and which benefits and risks they deemed most important.
  Arms: Electronic Patient Decision Aid
Behavioral: Standard Resource Sheet — Women allocated to the control intervention will login to the study website and receive a printable PDF containing references to standard published information on antidepressant use in pregnancy. This ensures women have access to accurate information on the benefits and risks of antidepressant medication in pregnancy (even though they will not receive the PDA).
  Women who are assigned the control condition AND who are not receiving care from Women's College Hospital Reproductive Life Stages Program will receive waitlisted access to the intervention after data collected at 4 weeks post-randomization.

SUMMARY:
The purpose of this pilot study is to examine the feasibility of conducting a multi-site randomized controlled trial whose aim will be to evaluate the effectiveness of a Patient Decision Aid (PDA) for antidepressant use in pregnancy.

DETAILED DESCRIPTION:
Depression in pregnancy is common, affecting up to 10% of women and represents serious risk to mother and infant. Unfortunately, antidepressant medication, a first-line treatment for depression in pregnancy, also comes with risks, making this a complex decision. Clinical care appears to be insufficient for ensuring that women make decisions that are consistent with their own values and with which they feel satisfied. Patient decision support tools can address such barriers. We have created a patient decision aid (PDA) that has the potential to improve the decision-making process for women regarding antidepressant use in pregnancy in conjunction with clinical care. The overall objective of this project is to inform the development of a larger, international RCT to assess the efficacy of our PDA for antidepressant use in pregnancy. To achieve this objective, we will assess the feasibility of our clinical trial protocol to evaluate the PDA and determine the preliminary effect size for a larger multi-site efficacy study. The primary outcome for this pilot study is the feasibility of conducting a large randomized controlled trial to evaluate the efficacy of the PDA. This includes feasibility (how well the trial protocol can be implemented), acceptability (usability and tolerability of the intervention) and adherence (the degree to which the trial protocol is followed). We hypothesize that our protocol will be feasible, that the PDA will have a high degree of acceptability, and that adherence to the protocol will be high.

ELIGIBILITY:
Inclusion criteria:

1. Are females aged >18 years old, and
2. Are either planning a pregnancy OR are <30 weeks gestation at enrollment, and
3. Have been offered to start or continue SSRI or SNRI anti-depressant medication as a treatment option for depression by their clinical provider at one of the study sites, and
4. Have moderate-to-high decisional conflict (score of >25 on the Decisional Conflict Scale)

Exclusion criteria:

1. Have had alcohol or substance abuse or dependence in the previous 12 months, or
2. Have active suicidal ideation or psychosis, or
3. Are incapable of consenting to participation, or
4. Have any major obstetrical complications or fetal cardiac anomaly in the current or in a past pregnancy (as this changes the risk/benefit ratio discussion in regards to antidepressant use), or
5. Are unable to read or unable to speak or understand English and do not have someone that can read the PDA to them, or
6. Have a visual impairment that would prevent them from being able to view the website.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-01; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | Up to one year from when the study starts enrolling participants
  Feasibility: Number of participants recruited into the study over Number of eligible patients

SECONDARY OUTCOMES:
Decisional Conflict Scale | Baseline (pre-randomization)
Knowledge about antidepressant treatment in pregnancy | Baseline (pre-randomization)
Edinburgh Postnatal Depression Scale | Baseline (pre-randomization)
Spielburg State-Trait Anxiety Inventory | Baseline (pre-randomization)
Edinburgh Postnatal Depression Scale | 4 Weeks post-randomization
Edinburgh Postnatal Depression Scale | 12 weeks postpartum (for participants who enrolled while pregnant) OR 6 months post-randomization (for women who enrolled while planning a pregnancy), only for participants who are seeing specialty psychiatric services
Spielburg State-Trait Anxiety Inventory | 4 Weeks post-randomization
Spielburg State-Trait Anxiety Inventory | 12 weeks postpartum (for participants who enrolled while pregnant) OR 6 months post-randomization (for women who enrolled while planning a pregnancy), only for participants who are seeing specialty psychiatric services
Decisional Conflict Scale | 4 Weeks post-randomization
Knowledge about antidepressant treatment in pregnancy | 4 Weeks post-randomization
PDA Acceptability Questionnaire | 4 Weeks post-randomization
Provider Perspective Survey | After all other participant data has been collected
Treatment Decision(s) | Baseline (pre-randomization)
Treatment Decision(s) | 4 Weeks post-randomization
Treatment Decision(s) | 12 weeks postpartum (for participants who enrolled while pregnant) OR 6 months post-randomization (for women who enrolled while planning a pregnancy), only for participants who are seeing specialty psychiatric services
Time between recruitment to first log-in to the study website | 4 weeks post-randomization
Self-reported satisfaction with the PDA by the participants | 4 Weeks post-randomization
Provider's perspective on the utility of the PDA in clinical practice | After all participant data has been collected
Study Website Usage | 4 Weeks post-randomization
  Composite measure comprised of: (1) number of participants who complete the PDA, (2) length of time required to complete the PDA, (3) number of log ins, (4) number of times the PDA is completed per participant, (5) total number of webpages viewed).
Number of participants who follow-up with their physician during the intended timeline | 4 weeks post-randomization, only for participants who are seeing specialty psychiatric services
The rate of follow-up data collection | 4 Weeks post-randomization
The rate of follow-up data collection | 12 weeks postpartum (for participants who enrolled while pregnant) OR 6 months post-randomization (for women who enrolled while planning a pregnancy), OR at 4 weeks post-randomization for women who are NOT seeing specialty perinatal psychiatry services

CONTACTS AND LOCATIONS:
Overall Officials: Simone Vigod, MD, MSc, Principal Investigator — Women's College Hospital
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vigod SN, Hussain-Shamsy N, Stewart DE, Grigoriadis S, Metcalfe K, Oberlander TF, Schram C, Taylor VH, Dennis CL. A patient decision aid for antidepressant use in pregnancy: Pilot randomized controlled trial. J Affect Disord. 2019 May 15;251:91-99. doi: 10.1016/j.jad.2019.01.051. Epub 2019 Mar 18. PMID 30913472
- [Derived] Vigod S, Hussain-Shamsy N, Grigoriadis S, Howard LM, Metcalfe K, Oberlander TF, Schram C, Stewart DE, Taylor VH, Dennis CL. A patient decision aid for antidepressant use in pregnancy: study protocol for a randomized controlled trial. Trials. 2016 Feb 29;17(1):110. doi: 10.1186/s13063-016-1233-4. PMID 26923796